CLINICAL TRIAL: NCT04841603
Title: Brief Digital CBT for Mood and Anxiety Symptoms in Acute Psychiatric Inpatients: a Randomized Feasibility Trial
Brief Title: Brief Digital CBT for Mood and Anxiety Symptoms in Acute Psychiatric Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Gaurav Sharma, Resident Physician, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116/2020-01
Record Dates: First submitted 2021-03-30; First posted 2021-04-12 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Anxiety; Depressive Symptoms; Distress, Emotional; Anxiety and Fear; Anxiety State; Mental Disorders, Severe; Psychiatric Hospitalization
Keywords: inpatient psychiatry; psychiatric admission; mobile app; inpatient CBT
MeSH Terms: conditions — Anxiety Disorders; Depression; Mental Disorders | interventions — Therapeutics; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): Treatment as usual
  Interventions: Device: Treatment as Usual
- Mindshift CBT (Experimental): Treatment as usual + Access to Mindshift CBT app
  Interventions: Device: Mindshift CBT

INTERVENTIONS:
Device: Mindshift CBT — A tablet with the Mindshift CBT app installed. Mindshift CBT is a free, evidence based app developed by Anxiety Canada, designed to help users reduce symptoms of anxiety and distress.
  Other Names: CBT mobile app
  Arms: Mindshift CBT
Device: Treatment as Usual — Treatment as usual. A tablet identical to the intervention group, but without the Mindshift CBT app is available for patients to use during their inpatient stay.
  Other Names: Tablet
  Arms: Treatment as usual

SUMMARY:
A randomized control trial examining the feasibility, acceptability, and preliminary efficacy of providing access to the MindShift CBT mobile app via tablet for acute psychiatric inpatients.

DETAILED DESCRIPTION:
Psychiatric inpatients expect more psychosocial intervention during their inpatient stay than they receive. During the COVID-19 pandemic, existing interventions have been further reduced. Mood and anxiety symptoms are common for all inpatients across diagnostic categories. Studies have shown that cognitive behavioural therapy (CBT) can be effective for treating these symptoms among inpatients. The purpose of this study is to determine whether the Mindshift CBT app (an app based on principles of cognitive behavioural therapy) is an acceptable, feasible, and useable intervention for inpatients.

The Mindshift CBT app is a tool designed and maintained by Anxiety Canada. It includes tools for daily mood check-ins, healthy thinking, calming intense emotions, and taking actions to change behaviours associated with anxiety and low mood. It also includes information about the common types of anxiety.

The proposed trial includes 12 patients per arm. All participants in control and intervention groups will have access to assigned tablet devices throughout the study period, though only those in the intervention group will have the MindShift CBT app on their device. All participants will undergo assessments at baseline and at the end of the intervention period (1 week).

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the acute inpatient unit
* Fluent in English
* Dynamic Appraisal for Situational Aggression (DASA) score <=3
* Capable to consent to participation as assessed by the treating physician

Exclusion Criteria:

* Diagnosis of moderate-severe learning disability
* Diagnosis of moderate-severe neurocognitive disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Retention rates | 1 week
  Feasibility - whether the intervention is possible in the acute inpatient setting
Recruitment rates | 1 week
  Feasibility - whether the intervention is possible in the acute inpatient setting
Client Satisfaction Questionnaire 8 (CSQ-8) | 1 week
  Acceptability - whether the intervention is appropriate for the acute inpatient setting. The CSQ-8 scores range from 8 to 32, with higher values indicating higher satisfaction with the intervention.
User Experience Questionnaire (UXQ) | 1 week
  Usability - whether the intervention is serviceable for its intended purpose. The UXQ has 11 items exploring characteristics informing usability of mobile apps, each scored from 0-10, for a total score ranging from 10-110 (with larger scores indicating increased usability).
Qualitative Data Analysis | 1 week
  From focus groups, to inform feasibility, usability, and acceptability

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | 1 week
  Preliminary efficacy - whether symptoms of depression are improved by the intervention. PHQ-9 is scored from 0 to 27 with higher scores indicating increasing severity of symptoms.
General Anxiety Disorder 7 Scale (GAD-7) | 1 week
  Preliminary efficacy - whether symptoms of anxiety are improved by the intervention. GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut points for mild, moderate, and severe anxiety.
Kessler Psychological Distress Scale (K10) | 1 week
  Preliminary efficacy - whether symptoms of distress are improved by the intervention. Scores range from 10 to 50, with increasing scores indicating increasing distress and severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ishrat Husain, MBBS, MD (Res.), MRCPsych, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Radcliffe J, Smith R. Acute in-patient psychiatry: how patients spend their time on acute psychiatric wards. Psychiatric Bulletin. 2007 May;31(5):167-70.
- [Background] Kösters M, Burlingame GM, Nachtigall C, Strauss B. A meta-analytic review of the effectiveness of inpatient group psychotherapy. Group Dynamics: Theory, Research, and Practice. 2006 Jun;10(2):146.
- [Background] Xia J, Merinder LB, Belgamwar MR. Psychoeducation for schizophrenia. Cochrane Database Syst Rev. 2011 Jun 15;2011(6):CD002831. doi: 10.1002/14651858.CD002831.pub2. PMID 21678337
- [Background] Cuijpers P, Clignet F, van Meijel B, van Straten A, Li J, Andersson G. Psychological treatment of depression in inpatients: a systematic review and meta-analysis. Clin Psychol Rev. 2011 Apr;31(3):353-60. doi: 10.1016/j.cpr.2011.01.002. Epub 2011 Jan 16. PMID 21382540
- [Background] Hopkins JE, Loeb SJ, Fick DM. Beyond satisfaction, what service users expect of inpatient mental health care: a literature review. J Psychiatr Ment Health Nurs. 2009 Dec;16(10):927-37. doi: 10.1111/j.1365-2850.2009.01501.x. PMID 19930367
- [Background] Paul AM, Fleming CJ. Anxiety management on campus: an evaluation of a mobile health intervention. J Technol Behav Sci 2018 Sep 19;4(1):58-61.
- [Background] Marshall JM, Dunstan DA, Bartik W. Effectiveness of Using Mental Health Mobile Apps as Digital Antidepressants for Reducing Anxiety and Depression: Protocol for a Multiple Baseline Across-Individuals Design. JMIR Res Protoc. 2020 Jul 5;9(7):e17159. doi: 10.2196/17159. PMID 32623368
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Husain MO et al. Evaluating the feasibility and acceptability of mobile health apps that deliver psychosocial interventions: using functional criteria to capture the user's experience (under review). Digital Health 2020.
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics: The Journal of Applied Statistics in the Pharmaceutical Industry. 2005 Oct;4(4):287-91.
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qualitative research in psychology. 2006 Jan 1;3(2):77-101.
- [Derived] Sharma G, Schlosser L, Jones BDM, Blumberger DM, Gratzer D, Husain MO, Mulsant BH, Rappaport L, Stergiopoulos V, Husain MI. Brief App-Based Cognitive Behavioral Therapy for Anxiety Symptoms in Psychiatric Inpatients: Feasibility Randomized Controlled Trial. JMIR Form Res. 2022 Nov 2;6(11):e38460. doi: 10.2196/38460. PMID 36322113